CLINICAL TRIAL: NCT03725891
Title: Comparison of Two Doses (81 mg Versus 162 mg) of Aspirin for the Prevention of Preeclampsia in Healthy, Nulliparous Obese and Overweight Pregnant Women: A Randomized Controlled Trial
Brief Title: Aspirin for Prevention of Preeclampsia in Healthy, Nulliparous Obese and Overweight Pregnant Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, hany farouk, Principal Investigator, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: aswu/196/7/18
Record Dates: First submitted 2018-10-29; First posted 2018-10-31 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Preeclampsia
Keywords: preeclampsia; low dose aspirin; high risk pregnancy
MeSH Terms: conditions — Pre-Eclampsia | interventions — Aspirin

STUDY DESIGN:
Intervention Model Description: This will be a randomized control trial to estimate the efficacy of two doses (81 mg versus 162 mg) of aspirin for prevention of preeclampsia in healthy, nulliparous obese and overweight pregnant women identified in the first trimester.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: both participants and researchers will be blinded to the intervention given
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aspirin 162 mg (Active Comparator): Aspirin 81mg tow tablet once a day from recruitment until 37 weeks or labor whichever comes first
  Interventions: Drug: Aspirin 162 mg
- Aspirin 81 mg plus placebo (Active Comparator): Aspirin 81mg one tablet once a day from recruitment until 37 weeks or labor whichever comes first plus placebo one tablet once a day from recruitment until 37 weeks or labor whichever comes first
  Interventions: Drug: Aspirin 81 mg; Drug: placebo

INTERVENTIONS:
Drug: Aspirin 162 mg — Aspirin 81mg two tablet once a day from recruitment until 37 weeks or labor whichever comes first
  Other Names: Active Comparator
  Arms: Aspirin 162 mg
Drug: Aspirin 81 mg — placebo one tablet once a day from recruitment until 37 weeks or labor whichever comes first
  Other Names: Active Comparator
  Arms: Aspirin 81 mg plus placebo
Drug: placebo — placebo one tablet once a day from recruitment until 37 weeks or labor whichever comes first
  Other Names: Active Comparator
  Arms: Aspirin 81 mg plus placebo

SUMMARY:
Preeclampsia is a pregnancy-specific syndrome that affects 3 - 5% of pregnancies. It is one of the main causes of maternal, fetal and neonatal morbidity and mortality, resulting in approximately 40,000 maternal deaths worldwide each year. Fortunately, preeclampsia-related deaths have been reduced remarkably in recent decades thanks to improvements in antenatal care and therapeutic interventions, and prophylactic use of low-dose aspirin in women who are at a higher risk of developing preeclampsia.

Effective prevention is rarely available for obstetric complications. Aspirin is one of them. Several meta-analyses456 suggested that aspirin prescription reduced the risk of preeclampsia and fetal growth restriction by 40-50% in an aspirin-dose-response pattern.

DETAILED DESCRIPTION:
Preterm preeclampsia is an important cause of maternal and perinatal death and complications. It is uncertain whether the intake of low-dose aspirin during pregnancy reduces the risk of preterm preeclampsia.

In a meta-analysis of individual-participant data from the trials, the effect of aspirin was not affected by the gestational age at the onset of therapy. In contrast, other meta-analyses showed that aspirin started at or before 16 weeks of gestation resulted in halving the rates of preeclampsia, fetal growth restriction, and perinatal death, whereas aspirin started after 16 weeks of gestation did not have a significant benefit. In addition, the beneficial effect of aspirin that was started at or before 16 weeks of gestation was dose-dependent, with a greater reduction in the incidence of preeclampsia being associated with a daily dose of aspirin of 100 mg or more.

This will be a randomized control trial to estimate the efficacy of two doses (81 mg versus 162 mg) of aspirin for prevention of preeclampsia in healthy, nulliparous obese and overweight pregnant women identified in the first trimester.

ELIGIBILITY:
Inclusion Criteria:

* healthy, nulliparous obese and overweight pregnant women identified in the first trimester.
* Give written informed consent.

Exclusion Criteria:

* Multiple gestations,
* fetal aneuploidy
* major fetal structural anomaly
* bleeding disorder
* allergy to aspirin
* women already on aspirin or heparin.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — This will be a randomized control trial to estimate the efficacy of two doses (81 mg versus 162 mg) of aspirin for prevention of preeclampsia in healthy, nulliparous obese and overweight pregnant women identified in the first trimester.
Enrollment: 600 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With early onset Preeclampsia | 6 months
  The number of cases of preeclampsia that appear in both groups before 34 weeks of pregnancy.Blood pressure greater than 140/90 on 2 occasions 6 hrs apart and significant proteinuria (greater than 300 mg in 24 hrs) before 34 weeks gestation

SECONDARY OUTCOMES:
Number of Participants With preeclampsia between 37 and 41 | 6 months
  The number of cases of preeclampsia that appear in both groups between 37 and 41 weeks of pregnancy
The number of cases of Fetal Growth Restriction | 6 months
  The number of cases of fetal growth restriction, defined as a fetal weight below the 10th percentile and an abnormal umbilical cord doppler that appear in both groups at any given time during pregnancy.
The number of cases of preterm birth | 6 months
  The number of cases delivered before 37 weeks gestation

CONTACTS AND LOCATIONS:
Overall Officials: hany f sallam, md, Principal Investigator — Aswan University Hospital
Locations (1):
- Aswan University, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: No